CLINICAL TRIAL: NCT00591240
Title: A Biochip for Rapid Diagnosis of Complicated Urinary Tract Infection
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B4872-R
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Urinary Tract Infections; Bladder, Neurogenic
Keywords: RNA, ribosomal, 16S; Biosensing techniques; Microchip analytical procedures
MeSH Terms: conditions — Urinary Tract Infections; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiplex pathogen identification.: Urine samples of patients at risk for urinary tract infections were collected. Biosensor based assays were used to detect the most common uropathogens in these samples. Analytical validity of the biosensor assays was examined by comparing biosensor results to those obtained using standard clinical microbiology laboratory methods. No interventions were performed.
- Antimicrobial susceptibility testing.: Urine samples of patients at risk of urinary tract infections were collected. Biosensor based antimicrobial susceptibility test, in concert with pathogen identification assay was directly performed on these samples. Analytical validity of the biosensor assays was examined by comparing biosensor results to those obtained using standard clinical microbiology laboratory methods. No interventions were performed.

SUMMARY:
The purpose of this proposal is clinical validation of an electrochemical biochip for rapid pathogen identification and antibiotic susceptibility determination.

DETAILED DESCRIPTION:
Point-of-care identification of pathogens and determination of antibiotic susceptibility will significantly improve the clinical management of urinary tract infection. We have previously developed a biochip based on microfabrication technology capable of rapid detection of pathogens. The specific objectives of the current proposal are: 1) Determination of microbial constituents in spinal cord injury (SCI) patients and development of additional species-specific probes against these pathogens; 2) Development of a rapid antibiotic susceptibility and molecular pyuria assay using the electrochemical biochip; and 3) Clinical validation of the biochip as a diagnostic test for urinary tract infection.

Within a single protocol, two non-interventional studies were conducted at different time points to achieve the aforementioned objectives. Sensitivity and specificity of the electrochemical biosensor based assay was demonstrated in each study.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected or at risk for complicated urinary tract infections

Exclusion Criteria:

* Gross contamination of urine samples at the time of collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at risk for urinary tract infections.
Sampling Method: Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Liao, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen CH, Lu Y, Sin ML, Mach KE, Zhang DD, Gau V, Liao JC, Wong PK. Antimicrobial susceptibility testing using high surface-to-volume ratio microchannels. Anal Chem. 2010 Feb 1;82(3):1012-9. doi: 10.1021/ac9022764. PMID 20055494
- [Result] Mach KE, Du CB, Phull H, Haake DA, Shih MC, Baron EJ, Liao JC. Multiplex pathogen identification for polymicrobial urinary tract infections using biosensor technology: a prospective clinical study. J Urol. 2009 Dec;182(6):2735-41. doi: 10.1016/j.juro.2009.08.028. Epub 2009 Oct 17. PMID 19837423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Urine samples were collected from participants at the Spinal Cord Injury Service at Veterans Affairs Palo Alto Health Care System for assay validation.
Groups:
- Multiplex Identification of Pathogens.: Urine samples of patients at risk for urinary tract infections were collected. Biosensor based assays were used to detect the most common uropathogens in these samples. Analytical validity of the biosensor assays was examined by comparing biosensor results to those obtained using standard clinical microbiology laboratory methods. No interventions were performed.
Period: Overall Study
Arm/Group | Multiplex Identification of Pathogens. | Antimicrobial Susceptibility Testing.
Started | 116 | 222
Completed | 116 | 222
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Research subjects recruited from spinal cord injury unit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiplex Identification of Pathogens. | Antimicrobial Susceptibility Testing. | Total
Number analyzed (Participants) | 116 | 222 | 338
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | NA — Age information was not collected for Group 2: Antimicrobial susceptibility testing. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | 100 | NA — Age information was not collected for Group 2: Antimicrobial susceptibility testing. | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | 16 | NA — Age information was not collected for Group 2: Antimicrobial susceptibility testing. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 112 | 215 | 327

OUTCOME MEASURES:

1. Primary Outcome: Clinical Validation of Biosensor Assays Used for Pathogen Identification and Antimicrobial Susceptibility Testing in Patients at Risk of Urinary Tract Infections.
Description: Study 1: Multiplex pathogen identification using biosensor based assay. We recruited 116 participants yielding 109 urine samples suitable for analysis and comparison between biosensor assays and standard urine culture. Biosensor based assays were used to detect multiple pathogens in the urine samples.
  Study 2: Antimicrobial susceptibility testing using biosensor based assay. We recruited 222 participants yielding 252 urine samples. Corresponding biosensor and clinical microbiology culture data was available for 215 samples. 73% (157) of these samples contained bacteria. Biosensor based antimicrobial susceptibility test, in concert with pathogen identification assay was directly performed on these samples.
Time Frame: Up to 1.5 years
Population: Urine samples were collected from participants at the Spinal Cord Injury Service for assay validation.
Measure: Number; unit: percentage of urine specimen
Units Other Than Participants: Urine specimen
Arm/Group | Multiplex Identification of Pathogens. | Antimicrobial Susceptibility Testing.
Number analyzed (Participants) | 116 | 222
Number analyzed (Urine specimen) | 109 | 157
percentage of urine specimen
  Biosensor sensitivity | 89 | 92
  Biosensor specificity | 100 | 97
  Negative predictive value | 76 | 81

ADVERSE EVENTS:
Description: Adverse events were not assessed as there were no interventions performed in these studies.
Arm/Group | Multiplex Identification of Pathogens. | Antimicrobial Susceptibility Testing.
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The trial is non-interventional. Future studies will focused on developing advanced prototypes with the option of using the biosensor platform to direct patient care in comparison with standard microbiology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No